CLINICAL TRIAL: NCT07235267
Title: Establishing the Reliability and Validity of Tele-Assessment for Functional Performance in Older Adults: A Comparative Study With Younger Individuals
Brief Title: Reliability and Validity of Tele-Assessment for Functional Performance in Older vs. Younger Adults
Status: Recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Sezen Karaborklu Argut, Dr., Assistant Professor, Istanbul University - Cerrahpasa
Other Study IDs: 2025.17031
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Older Adults (65 Years and Older); Geriatric Health; Young Adults

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary Cohort: Older Adults: Primary Cohort (Older adults) included individuals aged ≥65 years, living independently in the community, without severe cognitive, visual, or musculoskeletal impairments that would prevent participation.
- Comparison Cohort: Young Adults: Comparison Cohort (Young Adults) included healthy individuals aged 18-44 years, without acute or chronic health conditions affecting mobility.

SUMMARY:
This cross-sectional, comparative study aims to examine the intra-rater reliability, validity, and feasibility of tele-assessment versions of three functional mobility tests-the Timed Up and Go (TUG), 30-second Sit-to-Stand (30sSTS), and Gait Speed Test (GST)-in community-dwelling older adults (≥65 years). To provide a comparative perspective, the same assessments will also be administered to a younger, healthy control group (18-44 years). The study seeks to determine whether tele-assessment can serve as a robust and practical alternative to in-person testing, thereby enhancing accessibility and ensuring high-quality functional evaluation in geriatric populations.

ELIGIBILITY:
* Inclusion Criteria (Older Adults, ≥65 years) Community-dwelling Independent in activities of daily living Able to provide informed consent Capable of performing TUG, 30sSTS, and GST without assistance
* Inclusion Criteria (Younger Adults, 18-44 years) Healthy individuals without acute or chronic conditions affecting mobility Able to provide informed consent Capable of performing TUG, 30sSTS, and GST independently
* Exclusion Criteria (both groups) Diagnosed neurological disorders (other than age-related decline) Uncontrolled cardiovascular or metabolic disease Recent surgery or fractures Severe cognitive impairment Contraindications to physical activity Lack of access to required telecommunication technology

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Healthy Older Adults and Younger Adults (as control)
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go (TUG) | Baseline
  Time (seconds) to complete the test, assessed face-to-face and via tele-assessment.
Timed Up and Go (TUG) | One week later
  Time (seconds) to complete the test, assessed face-to-face and via tele-assessment.
30-second Sit-to-Stand Test (30sSTS) | Baseline
  Number of sit-to-stand repetitions performed within 30 seconds, assessed face-to-face and via tele-assessment.
30-second Sit-to-Stand Test (30sSTS) | One week later
  Number of sit-to-stand repetitions performed within 30 seconds, assessed face-to-face and via tele-assessment.
Gait Speed Test (GST) | Baseline
  Gait speed (m/s) over a 4-meter course, assessed face-to-face and via tele-assessment.
Gait Speed Test (GST) | One week later
  Gait speed (m/s) over a 4-meter course, assessed face-to-face and via tele-assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpaşa Faculty of Health Sciences, Istanbul, Buyukcekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided